CLINICAL TRIAL: NCT03736616
Title: Acalabrutinib Plus RICE for Patients With Relapsed/Refractory DLBCL Followed by Autologous Hematopoietic Cell Transplantation and Acalabrutinib Maintenance Therapy
Brief Title: Acalabrutinib Plus RICE for Relapsed/Refractory DLBCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Swedish Medical Center (Other)
Collaborators: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-LY-808-SCI
Record Dates: First submitted 2018-06-08; First posted 2018-11-09 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Carboplatin; Ifosfamide; Etoposide; Rituximab; Carmustine; Cytarabine; Melphalan; acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A: Transplant eligible (Experimental): Patients receive RICE: Rituximab 375mg/m2 IV d1, Ifosfamide 5000mg/m2, Carboplatin area under curve (AUC) 5 IV d2, Etoposide (VP16) 100mg/m2 IV d1-3 & Acalabrutinib 100mg oral BID d1-21. Cycle is 21 days for up to 3 cycles of treatment.
  BEAM chemotherapy & autoHSCT: BEAM given as Carmustine (BCNU) 300mg/m2 IV day -6 respective to stem cell infusion, VP16 200mg/m2 IV BID day -5 to day-2, Cytarabine (Ara-C) 200mg/m2 IV BID day -5 to day -2, and Melphalan 140mg/m2 IV day -1. Autologous hematopoietic stem cell infusion on day 0. Only patients with CR/PR after RICE acalabrutinib will undergo BEAM and autoHSCT
  Maintenance therapy: Post autoHSCT patients will receive Acalabrutinib 100mg oral BID starting on day +30 for 12 consecutive months or until progression or intolerance if occurs within those 12 months.
  Interventions: Drug: Carboplatin; Drug: Ifosfamide; Drug: Etoposide; Biological: Rituximab; Drug: Carmustine; Drug: Cytarabine; Drug: Melphalan; Other: Autologous HSCT; Drug: Acalabrutinib
- Cohort B: Transplant ineligible (Experimental): Patients receive RICE chemoimmunotherapy + Acalabrutinib Salvage therapy: RICE: Rituximab 375mg/m2 IV d1, Ifosfamide 5000mg/m2, Carboplatin AUC 5 IV d2, Etoposide 100mg/m2 IV d1-3. Acalabrutinib 100mg oral BID d1-21. Cycle is 21 days for up to 3 cycles of treatment.
  Maintenance therapy: Patients will receive Acalabrutinib 100mg oral BID for 12 consecutive months or until progression or intolerance if occurs within those 12 months. Maintenance therapy will only be given to patients with stable disease or better response after 3 cycles of RICE+ acalabrutinib
  Interventions: Drug: Carboplatin; Drug: Ifosfamide; Drug: Etoposide; Biological: Rituximab; Drug: Acalabrutinib

INTERVENTIONS:
Drug: Carboplatin — Chemotherapy
Drug: Ifosfamide — Chemotherapy
Drug: Etoposide — Chemotherapy
  Other Names: VP-16
Biological: Rituximab — Anti-CD20 mAb
  Other Names: Rituxan
Drug: Carmustine — Chemotherapy
  Other Names: BCNU
  Arms: Cohort A: Transplant eligible
Drug: Cytarabine — Chemotherapy
  Other Names: ARA-C
  Arms: Cohort A: Transplant eligible
Drug: Melphalan — Chemotherapy
  Arms: Cohort A: Transplant eligible
Other: Autologous HSCT — Cellular Therapy
  Other Names: Autologous Hematopoeitic Stem Cell Transplantation
  Arms: Cohort A: Transplant eligible
Drug: Acalabrutinib — Bruton's Tyrosine Kinase Inhibitor

SUMMARY:
To evaluate the tolerability,feasibility, and efficacy of combining acalabrutinib with RICE chemotherapy as second line therapy in relapsed/refractory DLBCL patients with separate primary objectives in each of in two cohorts:

Cohort A: Hematopoeitic stem cell transplantation (HSCT) eligible patients undergoing second-line salvage chemoimmunotherapy [Rituximab, Ifosfamide, Carboplatin, and Etoposide (RICE)] plus acalabrutinib:.

Cohort B: Individuals not eligible for HSCT undergoing second-line salvage chemoimmunotherapy [Rituximab, Ifosfamide, Carboplatin, and Etoposide (RICE)] plus acalabrutinib followed by acalabrutinib as a maintenance therapy

DETAILED DESCRIPTION:
This is a phase II study with a safety run-in. There will be two planned cohorts, Cohort A and Cohort B. Cohort A will be open to R/R DLBCL patients who are medically eligible for autologous HSCT (autoHSCT). Cohort B will be open to R/R DLBCL patients who are medically ineligible for autologous transplant. Historical outcomes from completed, published prospective clinical trials using RICE salvage chemotherapy will serve as a comparator population.

Safety run-in: To assess for safety of the combination of acalabrutinib and RICE chemotherapy, we will pause enrollment in both cohorts to assess for any safety concerns once a total 10 patients have been enrolled to either cohort. After the first ten patients have all completed at least one cycle of therapy without unacceptable or unexpected concerns, enrollment will resume. If there are concerns about adverse events or the ability of patients to proceed as expected to HSCT, then the study team will convene to determine whether the protocol should be modified. Data obtained for the first ten patients will be included in the data sample for final analysis.

Cohort A: After confirmation of medical eligibility for autologous HSCT, patients enrolled in Cohort A will receive 2 cycles of standard dose RICE salvage chemotherapy in combination with acalabrutinib 100mg twice daily (BID) day 1-21 of a 21 day cycle. After 2 cycles of therapy, patients will undergo autologous cell collection per standard institutional procedures. Acalabrutinib will be held 3 days before planned placement of an apheresis collection catheter and resumed 3 days after completion of stem cell collection and catheter removal. Patients will then receive a 3rd cycle of RICE chemotherapy in combination with acalabrutinib 100mg BID. For patients with bone marrow disease at enrollment, a repeat bone marrow will be performed after 2 cycles of salvage therapy, prior to autologous stem cell collection. For patients with continued bone marrow disease after 2 cycles of salvage therapy, a 3rd cycle may be given prior to autologous cell collection. PET-CT (PET3) will be performed 14-21 days after day 1 of cycle 3 to assess response. Those patients with complete response (CR) or partial response (PR) after PET3 will move onto autologous transplant with Carmustine, Etoposide, Cytarabine, and Melphalan (BEAM) conditioning within 28-42 days of PET3. After adequate hematopoietic recovery (expected around 30 days after autologous HSCT), patients will restart acalabrutinib 100mg BID as maintenance therapy for a period of 12 months. Patients with a minor response (MR) or stable disease (SD) after PET3 will delay HSCT and will continue acalabrutinib 100mg BID with repeat PET every 6 weeks. If patient converts to CR at subsequent PET-CT, they may proceed with BEAM autologous HSCT within 28-42 days of achieving this response followed by 12 months of post-transplant acalabrutinib maintenance. Patients with continued PR/MR/SD may continue on study, if felt to be clinically benefitting without limiting toxicity, but will not receive a transplant. Patients demonstrating progressive disease (PD) at any stage will be withdrawn from study treatment but their outcomes will be tracked and included in final data analysis.

Cohort B: Patients medically ineligible for autologous HSCT but fit for salvage chemotherapy will receive 3 cycles or RICE salvage chemotherapy in combination with acalabrutinib 100mg BID day 1-21 of a 21 day cycle followed by PET-CT (PET3) 14-21 days after start of Cycle 3. Patients with CR/PR/MR/SD would continue with acalabrutinib maintenance with repeat PET-CT every 3 months until disease progression or toxicity. Patients demonstrating progressive disease (PD) will be withdrawn from study treatment but their outcomes will be tracked and included in final data analysis.

Establishing the feasibility of combining acalabrutinib with RICE chemotherapy in transplant eligible and transplant ineligible patients with R/R DLBCL will provide the foundation for a larger study of efficacy and long-term outcomes of the combination therapy for patients with R/R DLBCL. Such a study, if demonstrative of improvements in the complete response rate to salvage therapy at PET3, could provide evidence to support a new standard of care of for patients with R/R DLBCL.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed R/R DLBCL (per 2008 WHO classification)

   1. GCB or ABC cell of origin (by IHC using Hans algorithim)
   2. Transformation from prior indolent NHL is permitted
2. Relapsed or refractory to 1 prior line of anthracycline containing chemoimmunotherapy considered a standard 1st line therapy for DLBCL. Acceptable 1st line regimens are R-CHOP, R-EPOCH, or R-HyperCVAD chemotherapy regimens. Treatment with prior radiotherapy is allowed.
3. ECOG Performance status 0-2
4. Expected life expectancy of at least 3 months
5. Age 18 years or older
6. Disease measurable by FDG-PET that meets iWNHL size criteria (>1.5cm in longest diameter for lymph node or nodal mass, or >1.0cm in longest diameter for extranodal disease)
7. For Cohort A, patients must meet institutional eligibility guidelines for autologous HCT and all of the following

   1. Ejection fraction >40% by ECHO or MUGA
   2. Pulmonary function testing with corrected DLCO >50% of predicted
   3. Charlson Comorbidity Index <6
8. For Cohort B, patients must be considered medically ineligible for autologous HCT by fulfilling one or more of following.

   1. Do not meet inclusion criteria 7a, 7b, or 7c
   2. Age >75
   3. Any chronic medical condition, treated or untreated, for which the anticipated risks of autologous HCT are deemed by the investigator to outweigh potential benefit of autologous HCT.
9. Women of childbearing potential (WOCBP): Must use highly effective method of birth control during acalabrutinib treatment as well as for 2 days after the last dose of acalabrutinib Highly effective forms of contraception are defined in Section F13.
10. Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty.
11. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local subject privacy regulations).

Exclusion Criteria:

1. Inadequate organ function, including the following

   1. Hematologic: ANC <1000/uL, PLT <50,000/uL, and hemoglobin <7.0g/dL. If the patient is known to have bone marrow involvement with cytopenias directly attributed to disease, eligibility may be permitted per investigator's discretion.
   2. Hepatic: Total bilirubin ≥ 2.0 x ULN unless bilirubin elevation is due to Gilbert's syndrome or of non-hepatic origin. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥ 3 x upper limit of normal (ULN)
   3. Renal: Estimated creatinine clearance of < 29 mL/min, calculated using the formula of Cockcroft and Gault [(140-Age) • Mass (kg)/(72 • creatinine mg/dL); multiply by 0.85 if female].
   4. GI: Malabsorption syndrome or gastrointestinal disease that limits oral absorption of medication
2. Prior history of autologous or allogeneic HCT
3. Any known contraindication to ifosfamide, etoposide, carboplatin, or rituximab
4. Active chronic hepatitis B infection, defined by positive Hep B DNA PCR.
5. Active chronic hepatitis C infection, defined by positive Hep C RNA PCR
6. Requires treatment with a strong CYP3A inhibitor/inducer
7. Any history of known significant bleeding diathesis
8. History of stroke or intracranial hemorrhage within 6 months before the first dose of study drug.
9. Pregnant or breastfeeding
10. Any uncontrolled active fungal, bacterial, or viral systemic infection that is untreated or not responsive to antimicrobial therapy.
11. Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of acalabrutinib, or put the study outcomes at undue risk.
12. Uncontrolled HIV/AIDS. Patients who are HIV positive, but clinically stable and compliant with HAART >3months and with CD4 >200 may be considered for eligibility at the investigators discretion unless taking excluded strong CYP3A inhibitor/inducer
13. Prior exposure to a BTK inhibitor
14. Prior malignancy (other than DLBCL or indolent NHL), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for ≥ 2 years or which will not limit survival to < 2 years. Note: these cases must be discussed with the principal investigator
15. Known central nervous system metastases and/or carcinomatous meningitis. Brain metastases, but not carcinomatous meningitis, are allowed if they had been previously treated (either surgically resected or by radiation therapy) and had remained stable by repeat imaging ≥ 4 weeks after treatment before enrolling on this protocol.
16. Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or corrected QT interval (QTc) > 500 msec at screening (By Fridericia's formula). Atrial fibrillation that is controlled or considered stable by the investigator is permitted.
17. Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening.
18. Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon) within 7 days of first dose of study drug.
19. Requires treatment with proton pump inhibitors (eg, omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study.
20. Major surgical procedure within 28 days of first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
21. Subject has received anti-cancer therapy within a period of 14 days or 5 half-lives (whichever is shorter) or radiotherapy within 28 days of first dose of study drug.
22. Concurrent participation in another therapeutic clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2019-08-16 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Cohort A: Complete Response Rate | 10 weeks
  To estimate the confirmed complete response (CR) rate (RECIL 2017 criteria) prior to transplant in patients undergoing second-line therapy for relapsed/refractory DLBCL.
Cohort B: Progression Free Survival | 1 year
  To estimate the one-year progression free survival rate in patients undergoing second-line induction and maintenance therapy for relapsed/refractory DLBCL.

SECONDARY OUTCOMES:
Cohort A: Treatment Response | 10 weeks
  To determine the proportion of patients who complete 3 cycles of acalabrutinib with RICE therapy and achieve treatment response sufficient to continue on to receive planned auto HCT.
Cohort B: Treatment Completion | 17 weeks
  To determine the proportion of patients in Cohort B who complete 3 cycles of acalabrutinib with RICE therapy and 2 cycles or more of maintenance acalabrutinib.

OTHER OUTCOMES:
Cohorts A and B: Overall Response Rate | 1 year
  To measure the overall response rate (ORR) at 1 year following study initiation
Cohorts A and B: Incidence of treatment-related Grade 3 and 4 Adverse events as assessed by CTCAE v4.0 | 1.5 years
  Evaluate incidence of grade 3 or grade 4 treatment related adverse events as assessed by CTCAE v4.0
Cohorts A and B: Incidence of Serious Adverse Events | 1.5 years
  Evaluate incidence of protocol defined serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Krish Patel, MD, Principal Investigator — Swedish Medical Center
Locations (1):
- Swedish Cancer Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No